CLINICAL TRIAL: NCT03131622
Title: Impact of Ibis, a Digital Health Solution for Patient Activation and Early Intervention, on Acute Care Utilization by Patients With Advanced COPD
Brief Title: Impact of Ibis on Patients With Advanced COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Senscio Systems (Industry)
Collaborators: Central Maine Medical Family (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Senscio-001
Record Dates: First submitted 2016-12-13; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Digital Therapeutics (Experimental): Patients assigned to the digital therapeutics arm will receive Ibis and all the associate services.
  Interventions: Behavioral: Digital Therapeutics
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Digital Therapeutics
  Arms: Digital Therapeutics

SUMMARY:
The purpose of this research is to determine if Ibis™, a digital therapeutics solution developed by Senscio Systems, reduces the emergency room visits and hospitalizations of patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Gold Stage II with a CAT Score above 19
* Gold Stage III/IV with a CAT Score above 14

Exclusion Criteria:

* Cognitive or physical impediments that inhibits patients from interacting with our digital therapeutics platform.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Acute Care Utilization | 6 months and then again at 1 year

IPD SHARING:
Plan to Share IPD: Undecided